CLINICAL TRIAL: NCT00909571
Title: A Phase 3 Pilot Study to Describe the Pharmacokinetics of Tacrolimus in Patients Undergoing Primary Liver Donor Liver Transplantation Treated With Prograf Injection and Modified Release Tacrolimus Based Immunosuppressive Regimen
Brief Title: Pharmacokinetics of Tacrolimus in Liver Transplantation Patients Treated With Prograf and Modified Release Tacrolimus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma Korea, Inc. (Industry)
Responsible Party: Director, Astellas Pharma, Inc
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: MR-08-04-KOR
Record Dates: First submitted 2009-05-27; First posted 2009-05-28 (Estimated); Last update posted 2010-04-16 (Estimated); Status verified 2010-04

CONDITIONS: Liver Transplantation
Keywords: FK506E; MR4; Prograf; Tacrolimus; Living Liver Transplantation
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1. FK506E high dose group (Experimental)
  Interventions: Drug: FK506E (modified release tacrolimus); Drug: Prograf (tacrolimus)
- 2. FK506E low dose group (Experimental)
  Interventions: Drug: FK506E (modified release tacrolimus); Drug: Prograf (tacrolimus)

INTERVENTIONS:
Drug: FK506E (modified release tacrolimus) — oral
  Other Names: MR4, modified release Tacrolimus
Drug: Prograf (tacrolimus) — injection
  Other Names: FK506; tacrolimus

SUMMARY:
Tacrolimus pharmacokinetics study in primary living donor liver transplantation patients with Tacrolimus based immunosuppressive regimens.

DETAILED DESCRIPTION:
To describe the pharmacokinetics of Tacrolimus when administered as two different doses of modified release formulation FK506E(MR4) combined with Prograf injection in patients undergoing primary living donor liver transplantation based on the single center (Asan Medical Center) standard protocol regimen.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving a primary partial liver graft from a living donor
* Patients must receive the first dose of Tacrolimus after surgery and are expected to be maintained on Tacrolimus throughout the study

Exclusion Criteria:

* Patients receiving a multi-organ transplantation or having previously received an organ transplantation
* Patients receiving an auxiliary graft or in whom a bio-artificial liver has been used
* Patients allergic or intolerant to macrolide antibodies or Tacrolimus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-04; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Assessment of pharmacokinetic parameters | Day 6 and Day 14

SECONDARY OUTCOMES:
Incidence of acute rejection | within 12 weeks
Time to acute rejection | within 12 weeks
Assessment of graft survival | within 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Korea, Inc.
Locations (1):
- Seoul, South Korea